CLINICAL TRIAL: NCT00657839
Title: A Randomized, Double-blind, Placebo-controlled, Multi-center, Parallel Group Study to Assess the Efficacy of Vardenafil in the Treatment of Subjects With Symptomatic Benign Prostatic Hyperplasia
Brief Title: Assessment of Efficacy of Vardenafil in the Treatment of Subjects With Symptomatic Benign Prostatic Hyperplasia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 11863; EudraCT No. 2005-002796-32
Record Dates: First submitted 2008-04-09; First posted 2008-04-14 (Estimated); Last update posted 2014-10-28 (Estimated); Status verified 2014-10

CONDITIONS: Benign Prostatic Hyperplasia
Keywords: Benign Prostate Hyperplasia; Vardenafil; Genital Disease; Male: Signs and symptoms of Benign Prostate Hyperplasia
MeSH Terms: conditions — Prostatic Hyperplasia; Genital Diseases | interventions — Vardenafil Dihydrochloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Experimental)
  Interventions: Drug: Levitra (Vardenafil, BAY38-9456)
- Arm 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Levitra (Vardenafil, BAY38-9456) — 10 mg Vardenafil bid
  Arms: Arm 1
Drug: Placebo — Matching placebo
  Arms: Arm 2

SUMMARY:
Assessment of efficacy of vardenafil in the treatment of subjects with symptomatic Benign Prostatic Hyperplasia.The purpose of this study is to find out whether vardenafil can improve the lower urinary tract symptoms of benign prostatic hyperplasia after 8 weeks of daily administration of 10 mg BID.

ELIGIBILITY:
Inclusion Criteria:

* Males 45 to 64 years of age
* Lower urinary tract symptoms > 6 months
* International Prostate Symptom Score > 12

Exclusion Criteria:

* Prostate Specific Antigen > 3 ng/ml
* Residual urine volume > 150 m
* History of myocardial infarction, stroke or life-threatening arrhythmia within the prior 6 months
* Nitrate use
* Other exclusion criteria apply acc. to Summary of Product Characteristics

Ages: 45 Years to 64 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 222 (Actual)
Dates: Start 2005-10; Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
International Prostate Symptom Score and maximal urinary flow | 8 weeks

SECONDARY OUTCOMES:
International Prostate Symptom Score, storing and voiding subscore | 8 weeks
IIEF-EF domains score | 8 weeks
Safety and tolerability | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (14):
- Germany (14):
  - Biberach, Baden-Württemberg / 277
  - München, Bayern / 280
  - Rosenheim, Bayern / 280
  - Starnberg, Bayern / 280
  - Weiden, Bayern / 280
  - Hamburg, Hamburg / 287
  - Marburg, Hessen / 307
  - Tostedt, Niedersachsen / 292
  - Osnabrück, Niedersachsen / 293
  - Düsseldorf, Nordrhein-Westfalen / 296
  - Leverkusen, Nordrhein-Westfalen / 331
  - Mülheim, Nordrhein-Westfalen / 481
  - Leipzig, Sachsen / 313
  - Kiel, Schleswig-Holstein / 306

REFERENCES:
- See also: Click here to find information about studies related to Bayer Healthcare products conducted in Europe — http://www.clinicaltrialsregister.eu/